CLINICAL TRIAL: NCT07356843
Title: Implementing Community Palliative Care for People With Heart Failure
Brief Title: Palliative Care for People With HF
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Lyndsay DeGroot, Assistant Professor Nursing, Indiana University
Other Study IDs: 28648
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Congestive Heart Failure; Congestive Heart Failure(CHF); Congestive Heart Failure (CHF); Congestive Heart Failure Chronic
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ADAPT — Concurrent mixed methods design with rapid qualitative analysis of data from semi-structured interviews, structured clinic observations, and descriptive analysis of surveys. Participants will include clinical providers (e.g. physicians, advanced practice providers, nurses, social workers), staff, and leadership at IU Health. As opposed to traditional qualitative methods, rapid qualitative approaches are commonly used in implementation-focused research to guide real-time implementation processes.13 Findings will identify potential clinical partnership site(s) and inform selection and tailoring of strategies to implement ADAPT in a partner clinical site in the next stage of this project.

SUMMARY:
Imagine having heart failure, a condition where the heart struggles to pump blood, making daily life hard. People with heart failure often don't feel well and end up going to the hospital a lot. Many of these people could feel better with extra help, but there aren't many programs that offer support beyond usual heart failure treatments. That's where the ADAPT program comes in, which stands for "Advancing Symptom Alleviation with Palliative Treatment." In this program, nurses and social workers call people weekly, helping them manage their toughest symptoms, offering tools to cope with heart failure, and keeping the patients' current doctors involved. We tested this program in a research study with heart failure patients and found that it improved their quality of life and lowered depression, anxiety, and heart failure symptoms. We now want to see if the ADAPT program will work in the community, outside of a research setting, so that more people could benefit from it. Specifically, we want to know: can the ADAPT program work well in new places? Will patients and their families find it helpful? Most importantly, can it help improve the lives of people with heart failure in these new settings? To answer these questions, I'll team up with healthcare providers to 1) ask how we can adjust the ADAPT program to work well in various settings (e.g. primary care, heart failure clinic) and 2) use this information to create simple materials and trainings to help them easily provide ADAPT. This will prepare us for the next phase of this project to test out the new ADAPT program.

ELIGIBILITY:
Inclusion Criteria:

Outpatient clinician or staff member with at least 6 months of experience caring for patients with HF (e.g. physician, physician assistant, nurse practitioner, registered nurse, social worker, psychologist, medical assistant) or healthcare leadership personnel (e.g. Chief Nursing Officer, Clinic Medical Director etc.) 18 years or older

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient clinician or staff member with at least 6 months of experience caring for patients with HF
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Qualitative Themes | Single time point interview and survey
  Qualitative themes from interviews and clinic observations and descriptive summary statistics (e.g. means, percentages) of barriers and facilitators from pCAT and PCSI surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Lyndsay DeGroot, PhD, RN, Principal Investigator — Indiana University School of Medicine
Locations (1):
- IUHealth, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
Qualitative interview data is often identifiable

REFERENCES:
- [Background] Fernandez ME, Ten Hoor GA, van Lieshout S, Rodriguez SA, Beidas RS, Parcel G, Ruiter RAC, Markham CM, Kok G. Implementation Mapping: Using Intervention Mapping to Develop Implementation Strategies. Front Public Health. 2019 Jun 18;7:158. doi: 10.3389/fpubh.2019.00158. eCollection 2019. PMID 31275915
- [Background] Powell BJ, Waltz TJ, Chinman MJ, Damschroder LJ, Smith JL, Matthieu MM, Proctor EK, Kirchner JE. A refined compilation of implementation strategies: results from the Expert Recommendations for Implementing Change (ERIC) project. Implement Sci. 2015 Feb 12;10:21. doi: 10.1186/s13012-015-0209-1. PMID 25889199
- [Background] Gertner AK, Franklin J, Roth I, Cruden GH, Haley AD, Finley EP, Hamilton AB, Palinkas LA, Powell BJ. A scoping review of the use of ethnographic approaches in implementation research and recommendations for reporting. Implement Res Pract. 2021 Jan-Dec;2:2633489521992743. doi: 10.1177/2633489521992743. Epub 2021 Mar 16. PMID 34056611
- [Background] Kowalski CP, Nevedal AL, Finley EP, Young JP, Lewinski AA, Midboe AM, Hamilton AB. Planning for and Assessing Rigor in Rapid Qualitative Analysis (PARRQA): a consensus-based framework for designing, conducting, and reporting. Implement Sci. 2024 Oct 11;19(1):71. doi: 10.1186/s13012-024-01397-1. PMID 39394597
- [Background] Keniston A, McBeth L, Astik G, Auerbach A, Busch J, Kangelaris KN, Kulkarni SA, Linker AS, Sakumoto M, Leykum L, Burden M. Practical Applications of Rapid Qualitative Analysis for Operations, Quality Improvement, and Research in Dynamically Changing Hospital Environments. Jt Comm J Qual Patient Saf. 2023 Feb;49(2):98-104. doi: 10.1016/j.jcjq.2022.11.003. Epub 2022 Nov 7. PMID 36585315
- [Background] Gale RC, Wu J, Erhardt T, Bounthavong M, Reardon CM, Damschroder LJ, Midboe AM. Comparison of rapid vs in-depth qualitative analytic methods from a process evaluation of academic detailing in the Veterans Health Administration. Implement Sci. 2019 Feb 1;14(1):11. doi: 10.1186/s13012-019-0853-y. PMID 30709368
- [Background] Vindrola-Padros C, Johnson GA. Rapid Techniques in Qualitative Research: A Critical Review of the Literature. Qual Health Res. 2020 Aug;30(10):1596-1604. doi: 10.1177/1049732320921835. PMID 32667277
- [Background] Feldstein AC, Glasgow RE. A practical, robust implementation and sustainability model (PRISM) for integrating research findings into practice. Jt Comm J Qual Patient Saf. 2008 Apr;34(4):228-43. doi: 10.1016/s1553-7250(08)34030-6. PMID 18468362
- [Background] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. BMJ. 2021 Sep 30;374:n2061. doi: 10.1136/bmj.n2061. PMID 34593508
- [Background] Nevedal AL, Reardon CM, Opra Widerquist MA, Jackson GL, Cutrona SL, White BS, Damschroder LJ. Rapid versus traditional qualitative analysis using the Consolidated Framework for Implementation Research (CFIR). Implement Sci. 2021 Jul 2;16(1):67. doi: 10.1186/s13012-021-01111-5. PMID 34215286
- [Background] Bekelman DB, Feser W, Morgan B, Welsh CH, Parsons EC, Paden G, Baron A, Hattler B, McBryde C, Cheng A, Lange AV, Au DH. Nurse and Social Worker Palliative Telecare Team and Quality of Life in Patients With COPD, Heart Failure, or Interstitial Lung Disease: The ADAPT Randomized Clinical Trial. JAMA. 2024 Jan 16;331(3):212-223. doi: 10.1001/jama.2023.24035. PMID 38227034
- [Background] Chyr LC, DeGroot L, Waldfogel JM, Hannum SM, Sloan DH, Cotter VT, Zhang A, Heughan JA, Wilson RF, Robinson KA, Dy SM. Implementation and Effectiveness of Integrating Palliative Care Into Ambulatory Care of Noncancer Serious Chronic Illness: Mixed Methods Review and Meta-Analysis. Ann Fam Med. 2022 Jan-Feb;20(1):77-83. doi: 10.1370/afm.2754. PMID 35074772
- [Background] Bekelman DB, Rabin BA, Nowels CT, Sahay A, Heidenreich PA, Fischer SM, Main DS. Barriers and Facilitators to Scaling Up Outpatient Palliative Care. J Palliat Med. 2016 Apr;19(4):456-9. doi: 10.1089/jpm.2015.0280. Epub 2016 Mar 14. PMID 26974489
- [Background] Gelfman LP, Blum M, Ogunniyi MO, McIlvennan CK, Kavalieratos D, Allen LA. Palliative Care Across the Spectrum of Heart Failure. JACC Heart Fail. 2024 Jun;12(6):973-989. doi: 10.1016/j.jchf.2024.01.010. Epub 2024 Mar 6. PMID 38456852
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499
- [Background] May P, Normand C, Cassel JB, Del Fabbro E, Fine RL, Menz R, Morrison CA, Penrod JD, Robinson C, Morrison RS. Economics of Palliative Care for Hospitalized Adults With Serious Illness: A Meta-analysis. JAMA Intern Med. 2018 Jun 1;178(6):820-829. doi: 10.1001/jamainternmed.2018.0750. PMID 29710177
- [Background] DeGroot L, Koirala B, Pavlovic N, Nelson K, Allen J, Davidson P, Abshire M. Outpatient Palliative Care in Heart Failure: An Integrative Review. J Palliat Med. 2020 Sep;23(9):1257-1269. doi: 10.1089/jpm.2020.0031. Epub 2020 Jun 9. PMID 32522132
- [Background] Diop MS, Rudolph JL, Zimmerman KM, Richter MA, Skarf LM. Palliative Care Interventions for Patients with Heart Failure: A Systematic Review and Meta-Analysis. J Palliat Med. 2017 Jan;20(1):84-92. doi: 10.1089/jpm.2016.0330. Epub 2016 Dec 2. PMID 27912043
- [Background] Kavalieratos D, Gelfman LP, Tycon LE, Riegel B, Bekelman DB, Ikejiani DZ, Goldstein N, Kimmel SE, Bakitas MA, Arnold RM. Palliative Care in Heart Failure: Rationale, Evidence, and Future Priorities. J Am Coll Cardiol. 2017 Oct 10;70(15):1919-1930. doi: 10.1016/j.jacc.2017.08.036. PMID 28982506
- [Background] Bozkurt B, Ahmad T, Alexander KM, Baker WL, Bosak K, Breathett K, Fonarow GC, Heidenreich P, Ho JE, Hsich E, Ibrahim NE, Jones LM, Khan SS, Khazanie P, Koelling T, Krumholz HM, Khush KK, Lee C, Morris AA, Page RL 2nd, Pandey A, Piano MR, Stehlik J, Stevenson LW, Teerlink JR, Vaduganathan M, Ziaeian B; Writing Committee Members. Heart Failure Epidemiology and Outcomes Statistics: A Report of the Heart Failure Society of America. J Card Fail. 2023 Oct;29(10):1412-1451. doi: 10.1016/j.cardfail.2023.07.006. Epub 2023 Sep 26. No abstract available. PMID 37797885
- [Background] DeGroot L, Pavlovic N, Perrin N, Gilotra NA, Dy SM, Davidson PM, Szanton SL, Saylor MA. Palliative Care Needs of Physically Frail Community-Dwelling Older Adults With Heart Failure. J Pain Symptom Manage. 2023 Jun;65(6):500-509. doi: 10.1016/j.jpainsymman.2023.01.016. Epub 2023 Feb 1. PMID 36736499
- [Background] DeGroot L, Pavlovic N, Perrin N, Gilotra NA, Miller H, Denfeld QE, McIlvennan CK, Dy SM, Davidson PM, Szanton SL, Abshire Saylor M. The Association of Unmet Palliative Care Needs and Physical Frailty With Clinical Outcomes: A Prospective Study of Adults With Heart Failure. J Cardiovasc Nurs. 2025 Jul-Aug 01;40(4):296-303. doi: 10.1097/JCN.0000000000001087. Epub 2024 Apr 17. PMID 38635901